CLINICAL TRIAL: NCT02651571
Title: Survival Rates of Patients With Mobile Bearing Total Knee Arthroplasty After 10 Years
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6267
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-01

CONDITIONS: Knee Replacement
Keywords: Knee; Replacement; Prosthesis; Mobile-bearing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The total knee replacement has become a routine procedure. Survival rate of over 90% after 10 years are generally reported. However, complications and reoperation may still occur for many reasons, and some of them may be related to component design: loosening (tibial above), polyethylene wear, knee stiffness, ligamentous instability, etc ... . Therefore, new designs can, at least in theory, improve the results of conventional models.

In this study, the investigators want to compare retrospectively data concerning survival rates of patients wearing total knee prosthesis with mobile plate for over 10 years, with the ones published in the literature for conventional fixed-bearing prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients wearing total knee prosthesis with mobile plate for over 10 years

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wearing total knee prosthesis with mobile plate for over 10 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Compare retrospectively data concerning survival rates of patients wearing total knee prosthesis with mobile plate for over 10 years, with the ones published in the literature for conventional fixed-bearing prostheses. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No